CLINICAL TRIAL: NCT06902402
Title: Evaluation of Safety and Efficacy of Three Flavors of Supportan® Drink in Cancer Patients in Taiwan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi Taiwan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Supp-015-CEN
Record Dates: First submitted 2025-03-12; First posted 2025-03-30 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Malnutrition (Calorie)
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportan® Drink (Experimental)
  Interventions: Dietary Supplement: Supportan® Drink, flavour Tropical Fruits; Dietary Supplement: Supportan® Drink, flavour Cappuccino; Dietary Supplement: Supportan® Drink, flavour Pineapple-Coconut

INTERVENTIONS:
Dietary Supplement: Supportan® Drink, flavour Tropical Fruits — flavour Tropical Fruits
Dietary Supplement: Supportan® Drink, flavour Cappuccino — flavour Cappuccino
Dietary Supplement: Supportan® Drink, flavour Pineapple-Coconut — flavour Pineapple-Coconut

SUMMARY:
The goal of this clinical trial is to demonstrate safety and efficacy of Supportan® Drink (three flavors:Tropical Fruits, Cappuccino, and Pineapple-Coconut), administered as oral nutritional supplement, that will be taken in addition to the patient's normal dietary intake to meet the daily nutritional targets. in cancer patients. The main questions it aims to answer are:

Primary Efficacy Endpoint 1. Change in body weight from Baseline to end of treatment at Week 4 (Week 4 -Baseline) Secondary Efficacy Endpoints

1. Change in CRP from Baseline to Week 2 and to end of treatment at Week 4 (Week 2 - Baseline, Week 4 -Baseline)

Participants will be enrolled in one of three flavor group by his/her recruiting time. Each subject needs visit hospital at baseline, week 2 and week 4 for checkups and test. And he/she needs take two bottles of Supportan Drink per day. During the study periods, subjects need write down his/her dietary records every day for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving chemotherapy and/or radiotherapy, or immunotherapy, or targeted therapy;
2. Patient with diagnosed cancer of any type (e.g., head and neck cancer, lung cancer, digestive tract cancer, breast cancer);
3. Patient with or at risk of malnutrition defined as meeting Malnutrition Universal Screening Tool (MUST) with score ≥2;
4. Capable of using oral nutritional supplementation;
5. Written informed consent from patient.

Exclusion Criteria:

1. Patient with documented diagnosis of liver, kidney or heart disease in the hospital's electronic medical record (EMR); severity of disease evaluated by Investigator as not being suitable to participate in this study;
2. Current alcohol or substance abuse as assessed by Investigator;
3. Patient had a stroke in the past year and is after Investigator assessment judged as not yet clinically stable at the time of screening;
4. Patients who are diagnosed with mental illness or depression assessed by the Investigator as too severe for being suitable to participate in this study;
5. Pregnant or breastfeeding woman;
6. Allergic to any ingredient of the investigational products;
7. Patients receiving or having received standard (not disease specific) oral nutritional supplements (ONS), standard enteral formula/tube feeding or standard parenteral cancerspecific nutrition supplements in the last 3 days;
8. Patients receiving or having received ONS, enteral formula/tube feeding or parenteral nutrition with high fish oil or high EPA/DHA content (above 1 g/day) in the last 28 days;
9. Current use of medication, food supplements or ONS containing more than 500 mg of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)/day or fish oil capsules/supplements containing more than 500 mg EPA and DHA/day at screening;
10. Transfusion of blood products within 1 week before screening;
11. Surgery scheduled during the trial;
12. Participation in other clinical trials using investigational drugs within 14 days before the start of the trial or during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-04-14 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from Baseline to end of treatment at Week 4 (Week 4 -Baseline) | 4 weeks

SECONDARY OUTCOMES:
Change in CRP from Baseline to Week 2 and to end of treatment at Week 4 (Week 2 - Baseline, Week 4 - Baseline). | 4 weeks
Change in body weight from Baseline to Week 2 (Week 2 - Baseline). | 2 weeks
Change in BMI from Baseline to Week 2 and to end of treatment at Week 4 (Week 2 - Baseline, Week 4 - Baseline). | 4 weeks
Change in calorie intake from Baseline to Week 2 and to end of treatment at Week 4 (Week 2 - Baseline, Week 4 - Baseline) using 3-day Dietary Records and additional intake of calories and protein from Supportan® Drink. | 4 weeks
Investigational product (IP) treatment compliance rate (%) calculated from patient IP diaries. | 4 weeks
Change in protein intake from Baseline to Week 2 and to end of treatment at Week 4 (Week 2 - Baseline, Week 4 - Baseline) using 3-day Dietary Records and additional intake of calories and protein from Supportan® Drink. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital-Lover's lake branch, Keelung, Taiwan, Taiwan